CLINICAL TRIAL: NCT04586738
Title: Comparative Clinical Trial on the Efficacy and Safety of Non-resorbable Uveoscleral Implant Associated With Absorbable Collagen Matrix vs Isolated Absorbable Collagen Matrix in Non-perforating Deep Sclerectomy in Glaucoma Surgery
Brief Title: Efficacy and Safety of Non-resorbable Uveoscleral Implant Versus Absorbable Collagen Matrix in Non-perforating Deep Sclerectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Implants in deep sclerectomy
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Evaluations will be done an outcome assessor that do not know the intervention group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-resorbable uveoscleral implant associated with absorbable collagen matrix (Other): non-perforating deep sclerectomy surgery with non-resorbable uveoscleral implant associated with absorbable collagen matrix
  Interventions: Procedure: non-perforating deep sclerectomy surgery
- Isolated absorbable collagen matrix implant (Other): non-perforating deep sclerectomy surgery with isolated absorbable collagen matrix implant
  Interventions: Procedure: non-perforating deep sclerectomy surgery

INTERVENTIONS:
Procedure: non-perforating deep sclerectomy surgery — Non-penetrating deep sclerectomy is a non-perforating filtration procedure used for the surgical treatment of medically uncontrolled open angle glaucoma.This surgery is performed to facilitate the outflow of aqueous humour from the anterior chamber to the subconjunctival space through a natural membrane (trabeculo-Descemet's window). This enables a more physiological reduction of intraocular pressure to be achieved.

SUMMARY:
The aim of the study is to evaluate and compare the hypotensive efficacy at 24 months between non-perforating deep sclerectomy surgery with non-resorbable uveoscleral implant associated with absorbable collagen matrix versus non-perforating deep sclerectomy surgery with isolated absorbable collagen matrix implant.

DETAILED DESCRIPTION:
The aim of this study is to evaluate and compare the hypotensive efficacy at 24 months between two implants in glaucoma surgery. Non-perforating deep sclerectomy surgery with non-resorbable uveoscleral implant associated with absorbable collagen matrix versus non-perforating deep sclerectomy surgery with isolated absorbable collagen matrix implant.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age
* Primary or secondary open-angle glaucoma
* High intraocular pressure (greater than or equal to 18mmHg) despite using maximum medical treatment
* Intolerance to medication.

Exclusion Criteria:

* Patients with previous glaucoma surgery
* Previous ocular surgery in the last 6 months
* Previous history of Laser trabeculoplasty in the last 12 months
* Moderate or severe diabetic retinopathy
* Active or recurrent eye disease (uveitis)
* Plateau iris
* Ocular neovascularization
* Aphakia
* Neovascular angle-closure glaucoma
* Previous history of intraocular or extraocular malignant neoplasm
* Pregnancy or lactation period, axial length> 26mm and <20mm
* Unwillingness for participating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of Intraocular pressure | 24 hours after surgery, 3 months, 12 months, 24 months
  Comparison of intraocular pressure measurements

SECONDARY OUTCOMES:
Number of adverse events | 24 hours after surgery, 3 months, 12 months, 24 months
  Adverse events spontaneous by subject (Safety and tolerability)

CONTACTS AND LOCATIONS:
Overall Officials: Jéssica Botella García, MD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (2):
- Spain (2):
  - Jéssica Botella García, Barcelona
  - Hospital Universitario Germans Trias i Pujol, Barcelona